CLINICAL TRIAL: NCT03924960
Title: Effectiveness of High-intensity Interval Training Combined With Resistance Training in Patients With Fibromyalgia
Brief Title: High-intensity Interval Training in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Tuğba Atan, Assoc. Prof., Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-KAEK-023
Record Dates: First submitted 2019-04-22; First posted 2019-04-23 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; functional capacity; aerobic exercise
MeSH Terms: conditions — Fibromyalgia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (Experimental): Participants in this group will perform a 20-25 minutes of aerobic exercise with a maximum capacity of 3-4 minutes (HRmax 80-95%) and active recovery for 3-4 minutes (HRmax 30-50%), five exercise sessions per week for 6 weeks.
  Interventions: Behavioral: High-intensity interval training
- Moderate-intensity continuous training (Active Comparator): Participants in this group will perform a 30-45 minute ergometric cycling exercise at 65-70% of the measured maximum heart rate (HRmax), five exercise sessions per week for 6 weeks.
  Interventions: Behavioral: Moderate-intensity continuous training
- Control (Other): Usual care control group
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: High-intensity interval training — Participants in this group will perform a 20-25 minutes of aerobic exercise with a maximum capacity of 3-4 minutes (HRmax 80-95%) and active recovery for 3-4 minutes (HRmax 30-50%), five exercise sessions per week for 6 weeks.
  Arms: High-intensity interval training
Behavioral: Moderate-intensity continuous training — Participants in this group will perform a 30-45 minute ergometric cycling exercise at 65-70% of the measured maximum heart rate (HRmax), five exercise sessions per week for 6 weeks.
  Arms: Moderate-intensity continuous training
Behavioral: Control — Usual care control group
  Arms: Control

SUMMARY:
Fibromyalgia is a common rheumatic disease characterized by widespread musculoskeletal pain, tenderness, fatigue, sleep disorders, cognitive and somatic complaints. Patients often suffer many somatic and psychological symptoms which contributes negative effect on the health- related quality of life, physical performance and physical activity. Recently, the European League Against Rheumatism presented evidence based recommendations for the management of the fibromyalgia. Accordingly, prompt diagnosis and patient education is required for optimal management. A graduated approach with the aim of improving health-related quality of life should be followed. It should focus ﬁrst on non-pharmacological modalities and the only "strong for" evidence-based recommendation was the use of aerobic and strengthening exercise. Aerobic exercise with moderate intensity (60 to 70% of age-adjusted predicted maximum heart rate (maxHR)) with a frequency of two or three times per week for at least 4 to 6 weeks for a reduction of symptoms is recommended in the management of fibromyalgia. Low-intensity aerobic exercise (<50 % maxHR) is founded ineffective. In recent years, high intensity interval training (HIIT) is used as popular instead of moderate intensity continuous exercise training (MICT) in cardiac rehabilitation units. It is found superior to moderate intensity exercise in improving cardiovascular fitness as increases maximal oxygen consumption (VO2max). The investigators hypothesis is that 6 weeks of five weekly sessions of HIIT will show superior effect reducing the impact of fibromyalgia and improving pain degree, functional capacity and health-related quality of life in women with fibromyalgia compared to MICT.

DETAILED DESCRIPTION:
Fibromyalgia is a common rheumatic disease characterized by widespread musculoskeletal pain, tenderness, fatigue, sleep disorders, cognitive and somatic complaints. Patients often suffer many somatic and psychological symptoms which contributes negative effect on the health- related quality of life, physical performance and physical activity. Recently, the European League Against Rheumatism presented evidence based recommendations for the management of the fibromyalgia. Accordingly, prompt diagnosis and patient education is required for optimal management. A graduated approach with the aim of improving health-related quality of life should be followed. Pharmacotherapy is only recommended for severe pain and sleep disturbances. It should focus ﬁrst on non-pharmacological modalities and the only "strong for" evidence-based recommendation was the use of aerobic and strengthening exercise. Aerobic exercise with moderate intensity (60 to 70% of age-adjusted predicted maximum heart rate (maxHR)) with a frequency of two or three times per week for at least 4 to 6 weeks for a reduction of symptoms is recommended in the management of fibromyalgia. Low-intensity aerobic exercise (<50 % maxHR) is founded ineffective. In recent years, high intensity interval training (HIIT) is used as popular instead of moderate intensity continuous exercise training (MICT) in cardiac rehabilitation units. It is found superior to moderate intensity exercise in improving cardiovascular fitness as increases maximal oxygen consumption (VO2max). While the moderate intensity continuous aerobic exercise program lasts 30 to 60 minutes, HIIT contains 4-6 cycles of 1-4 minutes with a maximum effort and lasts approximately 20 minutes in total. Therefore, another advantage of HIIT is the need for a shorter time to achieve similar or greater effects compared to MICT. The investigatorshypothesis is that 6 weeks of five weekly sessions of HIIT will show superior effect reducing the impact of fibromyalgia and improving pain degree, functional capacity and health-related quality of life in women with fibromyalgia compared to MICT. Therefore, the aim of this study is to assess the effects of HIIT versus MICT on pain, functional capacity and quality of life in women with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed according to the American College of Rheumatology 2016 diagnostic criteria for fibromyalgia.

Exclusion Criteria:

* History of comorbid inflammatory rheumatic/ connective tissue diseases
* History of cardiovascular or musculoskeletal problems that could prevent them to participate in an exercise program.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female sex
Enrollment: 55 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia impact questionnaire | 6 weeks
  The FIQ was designed to measure the health status of patients with fibromyalgia.

SECONDARY OUTCOMES:
Visual analogue scale | 6 weeks
  Pain intensity was measured with visual analogue scale (0-10mm) which is used to measure musculoskeletal pain with very good reliability and validity.
Short- form health survey 36 | 6 weeks
  Short- form health survey 36 contains 36 items which are used to evaluate the quality of life of patients with chronic pain. It measures eight different domains that address physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitation and mental health. The score of each domain ranges from 0 (worse quality of life) to 100 (best quality of life).
Cardiorespiratory fitness | 6 weeks
  A symptom-limited maximal cardiopulmonary exercise test performed on a cycle ergometer at baseline and following six-week exercise intervention to measure maximal oxygen consumption (VO2maximum) (ml/ kg/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Atan, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Rognmo O, Hetland E, Helgerud J, Hoff J, Slordahl SA. High intensity aerobic interval exercise is superior to moderate intensity exercise for increasing aerobic capacity in patients with coronary artery disease. Eur J Cardiovasc Prev Rehabil. 2004 Jun;11(3):216-22. doi: 10.1097/01.hjr.0000131677.96762.0c. PMID 15179103
- [Derived] Atan T, Karavelioglu Y. Effectiveness of High-Intensity Interval Training vs Moderate-Intensity Continuous Training in Patients With Fibromyalgia: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Nov;101(11):1865-1876. doi: 10.1016/j.apmr.2020.05.022. Epub 2020 Jun 22. PMID 32585169